CLINICAL TRIAL: NCT00936650
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Dose-Titration Study to Assess the Efficacy and Safety of Twice-Daily Dose Regimens of an Oral Calcimimetic Agent AMG 073 (Cinacalcet) in Primary Hyperparathyroidism (PHPT)
Brief Title: A Study to Assess the Efficacy and Safety of Twice-Daily Dose Regimens of an Oral Calcimimetic Agent AMG 073 (Cinacalcet) in Primary Hyperparathyroidism (PHPT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 990120
Record Dates: First submitted 2009-06-04; First posted 2009-07-10 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Hyperparathyroidism, Primary
Keywords: Hyperparathyroidism, Primary; cinacalcet
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- cinacalcet (Experimental)
  Interventions: Drug: cinacalcet
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Subjects were titrated to doses of 30, 40, or 50 mg BID every 4 weeks in a 12 week titration period, depending on their serum calcium concentration. The dose was kept constant for the ensuing 40 weeks except for dose reductions for hypocalcemia.
  Arms: placebo
Drug: cinacalcet — Subjects were titrated to doses of 30, 40, or 50 mg BID every 4 weeks in a 12 week titration period, depending on their serum calcium concentration. The dose was kept constant for the ensuing 40 weeks except for dose reductions for hypocalcemia.
  Arms: cinacalcet

SUMMARY:
This randomized, placebo-controlled study in patients with primary HPT was designed to evaluate the efficacy, safety, pharmacokinetics, and health-related quality of life (HRQOL) of AMG 073 when administered 2 times a day (BID). The study consisted of 3 phases: a 12-week dose-titration phase, a 12-week maintenance phase, and a 28-week follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age at screening
* Using, in the opinion of the principal investigator, effective contraceptive measures
* Plasma iPTH concentration > 45 pg/mL on at least 2 occasions at least 7 days apart during the 12 months preceding day 0 (at least 1 of these determinations should have been made during screening by the central lab) and serum calcium concentration > 10.3 mg/dL and ≤ 12.5 mg/dL on at least 2 occasions at least 7 days apart
* Acceptable renal function, with an estimated creatinine clearance > 50 mL/min as determined by the Cockroft and Gault equation
* Acceptable hepatic function, defined as serum aspartate aminotransferase, alanine aminotansferase, and total bilirubin ≤ 2 times the upper limit of normal according to the range provided by the central laboratory
* Laboratory test results within the central laboratory's normal range for hematology, urinalysis, and clinical chemistry parameters not mentioned specifically in other inclusion and exclusion criteria
* Chest x-ray within the previous 12 months without evidence of an active infectious, inflammatory, or malignant process
* Subject or legally acceptable representative gave informed consent for participation in the study

Exclusion Criteria:

* Unstable medical condition, defined as having been hospitalized within 30 days before day 0
* Pregnant or nursing
* Body habitus that precluded accurate DXA measurements
* Therapy within 21 days before day 0 with systemic glucocorticoids, lithium, tricyclic antidepressants with the exception of amitriptyline and nortryptiline, thioridazine, haloperidol, flecainide or other drugs with a narrow therapeutic index that are primarily metabolized by hepatic cytochrome P450 (CYP) 2D6, drugs that affect renal tubular calcium handling (eg, thiazide or loop diuretics), or calcitonin
* Received, within 90 days before day 0, therapy with bisphosphonates, with fluoride, or changes in thyroid replacement therapy
* Dose changes in selective estrogen receptor modulators (SERMs), or significant changes in doses of estrogen within 90 days before day 0. If a subject had discontinued estrogen or SERM therapy, they must have been off treatment for at least 90 days before day 0
* Alcohol abuse, or use of illicit drugs, within 12 months before day 0
* Myocardial infarction (MI) within 6 months before day 0
* Ventricular rhythm disturbance requiring current treatment
* Seizures within 12 months before day 0
* History (within 5 years) of malignancy of any type, other than nonmelanomatous skin cancers or in situ cervical cancer
* Within the past 5 years, evidence of treatment for and/or active sarcoidosis, tuberculosis, or other diseases known to cause hypercalcemia
* History of familial hypocalciuric hypercalcemia (FHH)
* Uncontrolled diabetes, as defined by hemoglobin A1c (HbA1c) ≥ 8.0
* Gastrointestinal disorder that might have been associated with impaired absorption of orally dministered medications
* Inability to swallow tablets
* Known sensitivity to any of the products to be administered during the study
* Psychiatric disorder that would have interfered with understanding and giving informed consent or compliance with protocol requirements
* Other condition that might have reduced the chance of obtaining data (eg, known poor compliance) required by the protocol or that might have compromised the ability to give truly informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 1999-11; Primary Completion 2001-03 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with the mean of the maintenance phase serum calcium measurements ≤ 10.3 mg/dL and with a mean decrease of at least 0.5 mg/dL | 24 weeks

SECONDARY OUTCOMES:
The change from baseline and percent change from baseline in maintenance phase mean for the following variables: serum BALP, serum 1,25(OH)2D3, serum NTx, serum phosphorus, urinary calcium/creatinine ratio, urinary DPD/creatinine ratio, and urinary NTx/c | 24 weeks
The internal consistency reliability, discriminant validity, criterion validity, and responsiveness of the Medical Outcomes Short Form-36 (SF-36), Brief Symptom Inventory (BSI), and Visual Analogue Scale (VAS) | 52 weeks
Change from baseline in serum calcium, percent change from baseline in serum calcium, and the proportion of subjects maintaining a 12-week maintenance phase mean reduction of serum calcium from baseline of at least 0.5 mg/dL | 24 weeks
Change from baseline in iPTH, percent change from baseline in PTH, the proportion with baseline > 65 pg/mL who decrease to ≤ 65 pg/mL, and the proportion of all subjects with iPTH ≤ 65 pg/mL | 24 weeks
The percent change from baseline in BMD at weeks 24 and 52 as assessed by DXA scans of proximal femur (total femur and femoral neck), lumbar spine (L1-L4), forearm (ultra distal radius and 1/3 radius), and total body | 52 weeks
The pharmacokinetic profile of AMG 073 as determined with population-based methods | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Peacock M, Bilezikian JP, Klassen PS, Guo MD, Turner SA, Shoback D. Cinacalcet hydrochloride maintains long-term normocalcemia in patients with primary hyperparathyroidism. J Clin Endocrinol Metab. 2005 Jan;90(1):135-41. doi: 10.1210/jc.2004-0842. Epub 2004 Nov 2. PMID 15522938
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com